CLINICAL TRIAL: NCT00463749
Title: Trial to Compare Infarct Size and Occurrence of Contrast Dye Induced Nephropathy in Patients With Primary Percutaneous PCI in STEMI
Brief Title: Myocardial Salvage and Contrast Dye Induced Nephropathy Reduction by N-Acetylcystein
Acronym: LIPSIA-N-ACC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Holger Thiele, MD, University of Leipzig - Heart Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1111/2006
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-07

CONDITIONS: Myocardial Infarction
Keywords: primary PCI; nephropathy; infarct size; infarction; ST-elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Kidney Diseases; Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): High-dose N-Acetylcystein during percutaneous coronary intervention and for 2 days post intervention 2 x/day
  Interventions: Drug: Acetylcystein
- 2 (Placebo Comparator): Placebo (NaCl)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylcystein — high-dose N-Acetylcystein during PCI and for 2/day for 2 days
  Arms: 1
Drug: Placebo — NaCl as placebo
  Arms: 2

SUMMARY:
Acetylcystein is a potent antioxidans which is able to prevent contrast dye induced nephropathy in stable patients undergoing additional hydration.

In primary percutaneous intervention for infarction hydration is not possible. Therefore Acetylcystein might prevent contrast dye induced nephropathy.

Furthermore, it might reduce infarct size as a result of its antioxidant properties.

Clinical trials are missing so far examining the effects of Acetylcystein on nephropathy and infarct size.

ELIGIBILITY:
Inclusion Criteria:

* ST-elevation infarction (<12 hours)
* Angina

Exclusion Criteria:

* Prior fibrinolysis
* Dialysis
* Pregnancy
* Lactase-reduction
* Glucose-galactose malabsorption
* Known allergy to acetylcystein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage measured by magnetic resonance imaging | 4 days
prevention of nephropathy | 3 days

SECONDARY OUTCOMES:
ST-segment resolution | 90 min
TIMI flow | minutes
composite clinical endpoint (death, reinfarction, congestive heart failure) | 30 days
need for dialysis | 4 days
microvascular obstruction measured by magnetic resonance | 4 days
infarct size measured by magnetic resonance | 4 days
oxidative stress | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Study Chair — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] de Waha S, Eitel I, Desch S, Fuernau G, Lurz P, Stiermaier T, Blazek S, Schuler G, Thiele H. Prognosis after ST-elevation myocardial infarction: a study on cardiac magnetic resonance imaging versus clinical routine. Trials. 2014 Jun 25;15:249. doi: 10.1186/1745-6215-15-249. PMID 24962156
- [Derived] Fuernau G, Zaehringer S, Eitel I, de Waha S, Droppa M, Desch S, Schuler G, Adams V, Thiele H. Osteoprotegerin in ST-elevation myocardial infarction: prognostic impact and association with markers of myocardial damage by magnetic resonance imaging. Int J Cardiol. 2013 Sep 1;167(5):2134-9. doi: 10.1016/j.ijcard.2012.05.101. Epub 2012 Jun 15. PMID 22704876
- [Derived] Fuernau G, Eitel I, Franke V, Hildebrandt L, Meissner J, de Waha S, Lurz P, Gutberlet M, Desch S, Schuler G, Thiele H. Myocardium at risk in ST-segment elevation myocardial infarction comparison of T2-weighted edema imaging with the MR-assessed endocardial surface area and validation against angiographic scoring. JACC Cardiovasc Imaging. 2011 Sep;4(9):967-76. doi: 10.1016/j.jcmg.2011.02.023. PMID 21920334
- [Derived] Droppa M, Desch S, Blase P, Eitel I, Fuernau G, Schuler G, Adams V, Thiele H. Impact of N-acetylcysteine on contrast-induced nephropathy defined by cystatin C in patients with ST-elevation myocardial infarction undergoing primary angioplasty. Clin Res Cardiol. 2011 Nov;100(11):1037-43. doi: 10.1007/s00392-011-0338-8. Epub 2011 Jun 28. PMID 21710343
- [Derived] Eitel I, Blase P, Adams V, Hildebrand L, Desch S, Schuler G, Thiele H. Growth-differentiation factor 15 as predictor of mortality in acute reperfused ST-elevation myocardial infarction: insights from cardiovascular magnetic resonance. Heart. 2011 Apr;97(8):632-40. doi: 10.1136/hrt.2010.219543. Epub 2011 Feb 22. PMID 21345844
- [Derived] Thiele H, Hildebrand L, Schirdewahn C, Eitel I, Adams V, Fuernau G, Erbs S, Linke A, Diederich KW, Nowak M, Desch S, Gutberlet M, Schuler G. Impact of high-dose N-acetylcysteine versus placebo on contrast-induced nephropathy and myocardial reperfusion injury in unselected patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. The LIPSIA-N-ACC (Prospective, Single-Blind, Placebo-Controlled, Randomized Leipzig Immediate PercutaneouS Coronary Intervention Acute Myocardial Infarction N-ACC) Trial. J Am Coll Cardiol. 2010 May 18;55(20):2201-9. doi: 10.1016/j.jacc.2009.08.091. PMID 20466200
- [Derived] Eitel I, Nowak M, Stehl C, Adams V, Fuernau G, Hildebrand L, Desch S, Schuler G, Thiele H. Endothelin-1 release in acute myocardial infarction as a predictor of long-term prognosis and no-reflow assessed by contrast-enhanced magnetic resonance imaging. Am Heart J. 2010 May;159(5):882-90. doi: 10.1016/j.ahj.2010.02.019. PMID 20435200